CLINICAL TRIAL: NCT03289377
Title: NRC: Improving Healthcare for Cognitively Impaired Elders and Their Caregivers
Brief Title: NRC:Improving Healthcare for Cognitively Impaired Elders and Their Caregivers
Acronym: RDAD&APNs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Linda Teri, Professor, School of Nursing, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003731
Record Dates: First submitted 2017-09-14; First posted 2017-09-21 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Alzheimer Disease; Nurse Training
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RDAD training to APNs (Experimental): Half-day workshop to provide APNs with all skills necessary to conduct RDAD in their clinical settings. A subset of the trained APNs will implement RDAD as part of their ongoing care of persons with ADRD.
  Interventions: Behavioral: RDAD Training

INTERVENTIONS:
Behavioral: RDAD Training — An interactive processes of lecture, role-play, and discussion, APNs will have the opportunity to dissect all phases of RDAD to insure they understand the objectives, can enact the program, and feel confident they can problem-solve situations that arise. APNs will receive materials to insure they are knowledgeable about ADRD symptoms, behavior management techniques, and exercise safety.

SUMMARY:
An multi-stage mixed-method design will be employed to obtain both qualitative and quantitative data to address two study aims: (1) Evaluate and refine the delivery Reducing Disabilities in Alzheimer's Disease (RD- AD) training to advanced practice nurses and (2) Evaluate and refine the implementation of RD-AD by advanced practice nurses in their medical settings.

DETAILED DESCRIPTION:
Two waves of APNs (25 each wave/total 50) will receive RDAD training and be queried pre and post- training using both qualitative and quantitative procedures to determine: (1) Is RDAD training successfully received by advanced practice nurses? (2) Do they report it as relevant to improving the care they deliver to persons with Alzheimer's Disease and Related Dementias (ADRD)? (3) Does RDAD training of advanced practice nurses improve their level of knowledge about ADRD, their skills in providing ADRD care, and their level of confidence in providing this care?

A subset of advanced practice nurses (5 per wave, total of 10) will be recruited to implement RDAD as part of their ongoing care of persons with ADRD.

ELIGIBILITY:
Inclusion Criteria:

* Licensed by the Washington state Department of Health as an Advanced Registered Nurse Practitioner (ARNP),
* Hold a board certification as a Gerontological Nurse Practitioner, Adult Nurse Practitioner, or Family Nurse Practitioner,
* Work at least half time (0.50 FTE) in a clinical setting (primary care, internal medicine, sub-specialty, medical home), with a panel consisting of over 25% of patients over 65 years of age,
* Have no expectation for termination over the course of the study; and
* Agree to participate in all phases of the RDAD translational program.

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Physician Confidence in Dementia Care Skills | Change from baseline score at 2 months
  A 12-item self-report measure (administered to ARNPs) designed to measure perception of ability to address the care needs of patients with ADRD.
Sense of Competence in Dementia | Change from baseline score at 2 months
  A 17-item questionnaire covering 4 domains: job satisfaction, attitude towards dementia, work experience, and level of dementia knowledge.
Dementia Attitudes Scale | Change from baseline score at 2 months
  A 20-item scale to measures attitudes towards dementia with a two-factor structure; "dementia knowledge" and "social comfort".

SECONDARY OUTCOMES:
Focus Group Questions | At 2 months
  Questions to determine satisfaction with a acceptability of RDAD
Implementation Questions | At 2 months
  Questions to determine Acceptability of RDAD

CONTACTS AND LOCATIONS:
Overall Officials: Linda Teri, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teri L, Gibbons LE, McCurry SM, Logsdon RG, Buchner DM, Barlow WE, Kukull WA, LaCroix AZ, McCormick W, Larson EB. Exercise plus behavioral management in patients with Alzheimer disease: a randomized controlled trial. JAMA. 2003 Oct 15;290(15):2015-22. doi: 10.1001/jama.290.15.2015. PMID 14559955
- [Background] Brodaty H, Arasaratnam C. Meta-analysis of nonpharmacological interventions for neuropsychiatric symptoms of dementia. Am J Psychiatry. 2012 Sep;169(9):946-53. doi: 10.1176/appi.ajp.2012.11101529. PMID 22952073
- [Background] Small GW, Rabins PV, Barry PP, Buckholtz NS, DeKosky ST, Ferris SH, Finkel SI, Gwyther LP, Khachaturian ZS, Lebowitz BD, McRae TD, Morris JC, Oakley F, Schneider LS, Streim JE, Sunderland T, Teri LA, Tune LE. Diagnosis and treatment of Alzheimer disease and related disorders. Consensus statement of the American Association for Geriatric Psychiatry, the Alzheimer's Association, and the American Geriatrics Society. JAMA. 1997 Oct 22-29;278(16):1363-71. PMID 9343469
- [Background] Koch T, Iliffe S; Evidem Programme. The role of primary care in the recognition of and response to dementia. J Nutr Health Aging. 2010 Feb;14(2):107-9. doi: 10.1007/s12603-010-0021-1. No abstract available. PMID 20126958
- [Background] Kukull WA, Higdon R, Bowen JD, McCormick WC, Teri L, Schellenberg GD, van Belle G, Jolley L, Larson EB. Dementia and Alzheimer disease incidence: a prospective cohort study. Arch Neurol. 2002 Nov;59(11):1737-46. doi: 10.1001/archneur.59.11.1737. PMID 12433261
- [Background] Bruce DG, Paley GA, Nichols P, Roberts D, Underwood PJ, Schaper F. Physical disability contributes to caregiver stress in dementia caregivers. J Gerontol A Biol Sci Med Sci. 2005 Mar;60(3):345-9. doi: 10.1093/gerona/60.3.345. PMID 15860472
- [Background] Mohamed S, Rosenheck R, Lyketsos CG, Schneider LS. Caregiver burden in Alzheimer disease: cross-sectional and longitudinal patient correlates. Am J Geriatr Psychiatry. 2010 Oct;18(10):917-27. doi: 10.1097/JGP.0b013e3181d5745d. PMID 20808108
- [Background] Tun SM, Murman DL, Colenda CC. Concurrent validity of neuropsychiatric subgroups on caregiver burden in Alzheimer disease patients. Am J Geriatr Psychiatry. 2008 Jul;16(7):594-602. doi: 10.1097/JGP.0b013e318173f5fc. PMID 18591579
- [Background] Gaugler JE, Duval S, Anderson KA, Kane RL. Predicting nursing home admission in the U.S: a meta-analysis. BMC Geriatr. 2007 Jun 19;7:13. doi: 10.1186/1471-2318-7-13. PMID 17578574
- See also: Dementia and its implications for public health 2006 — http://www.cdc.gov/pcd/issues/2006/apr/05_0167.htm